CLINICAL TRIAL: NCT04963881
Title: Clinical Features and Pattern of Antiphospholipid Antibodies in Patients of Antiphospholipid Syndrome (APS) With Systemic Lupus Erythematosus (SLE).
Brief Title: Antiphospholipid Antibodies in Patients of Antiphospholipid Syndrome (APS) With Systemic Lupus Erythematosus (SLE).
Status: Completed | Type: Observational
Sponsor: Fatima Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheharbano Imran, Assistant Professor, Fatima Memorial Hospital
Other Study IDs: FMHCMD
Record Dates: First submitted 2021-06-18; First posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Anti-phospholipid Antibobodies in Patients of SLE Presenting With Thrombosis or Pregnancy Complications
Keywords: APLS, Thrombosis, antiphosphoilipid antibodies
MeSH Terms: conditions — Pregnancy Complications; Thrombosis | interventions — Antibody Formation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Antibody testing — Blood samples were taken and analyzed for APS antibodies

SUMMARY:
Evaluation of antiphospholipid antibodies (aPL) profile in Systemic lupus erythematosus (SLE) patients with obstetric and thrombotic complications.

Blood sample of the patients were taken for Anti-beta-2-glycoprotein 1(anti-b2GPI), anticardiolipin (aCL) and will be analyzed on Alegria based on ELISA.

DETAILED DESCRIPTION:
Antiphospholipid syndrome (APS) is characterized by presence of specific antiphospholipid antibodies (aPL) with history of thrombosis and/or pregnancy morbidity.

Anti-phospholipid antibodies (aPL) is a comprehensive antibody profile which includes lupus anticoagulant [LA], anticardiolipin antibodies [aCL], and/or anti-β2-glycoprotein-I antibodies [aβ2GPI]). A comprehensive antibody profile is needed for both diagnosis and classification of patients with APS, most significantly for the risk assessment of both pregnancy morbidity and thrombosis.

Double positivity (LA, aβ2GPI or ACL +) and triple positivity (LA, aβ2GPI+, ACL +) may have worse outcome and the patients with double and triple positivity may have recurrent thrombotic events.

Early detection of aPL antibodies may avert patients with many complication associated with SLE as well as from major thrombotic events because the detection of aPL in SLE has been proposed as a predictive and specific tool for the diagnosis of APLS in SLE.

aPL profile in SLE patients with obstetric and thrombotic complications was analyzed, to see the association of different anti phospholipid antibodies with different clinical features of APLS in SLE patients.

ELIGIBILITY:
Inclusion Criteria: Diagnosed patients of SLE presenting with thrombosis & pregnancy complication were studied

-

Exclusion Criteria:

* Patients of SLE without thrombosis

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients of SLE, both genders, presenting with thrombosis or pregnancy complications were studied.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
aPLS antibodies of any type and number lead to cumulative obstetric and thrombotic complication in patients of SLE. | 2 years
B2 GPI is more prevalent in patients with antiphospholipid syndrome | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fatima Memorial Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No